CLINICAL TRIAL: NCT06210672
Title: A Prospective Longitudinal Study of Natural History and Functional Status of Patients With Gamma-sarcoglycanopathy (LGMDR5)
Brief Title: Natural History Study in Patients With LGMDR5/2c
Status: Withdrawn | Type: Observational
Why Stopped: lack of financing
Sponsor: Atamyo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ATA-002-GSAR
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Gamma-sarcoglycanopathy
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, longitudinal, interventional, multicenter natural history study to better understand the LGMDR5/2c disease physiopathology. The duration of participation for each patient will be up to 24 months.

DETAILED DESCRIPTION:
Study duration Duration from First visit of first patient (FPFV) to Last visit of last patient (LPLV) : 3 years. Each patient will have a visit every 6 months over 2 years (5 visits in total).

Study primary objective is to characterize the disease course in gamma-sarcoglycanopathy (LGMDr5/2c) patients using standardized and disease appropriate evaluations.

Secondary objectives are to identify clinical, imaging and/or laboratory parameters that are indicators of the disease course in LGMD2c and to identify the best outcome measure for further therapeutics approaches

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 6 to less than 35 years of age
* Ambulant patients should be less than 12 years of age and able to walk/run 10 meters (item 29 of NSAD) in less than 15 sec
* Confirmed diagnosis of LGMDR5 (genotyping)
* FVC > 40%

Exclusion Criteria:

* Subjects with co-morbidity which may interfere with LGMDR5 natural evolution and/or evaluation of outcome measures
* Need of non-invasive ventilation > 16h per 24h or any invasive ventilation
* Left ventricular ejection fraction (LVEF) < 30% or prior heart failure decompensation requiring hospitalization
* Past participation in a gene therapy or cell therapy trial

Ages: 6 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study will enroll 30 ambulant pediatric patients less than 12 years of age (cohort 1) and 20 non-ambulant adolescent or young adults less than 35 years of age (cohort 2)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
North Star Assessment for Neuromuscular Disorders (NSAD) | Baseline through 24 months
  Change from baseline in NSAD score (with a score range from 0 to 54, the higher the score the better the ability)
Performance of Upper Limb (PUL) | Baseline through 24 months
  Change from baseline in PUL score (with a score range from 0 to 42, the higher the score the better the ability)
Timed Up and Go (TUG) | Baseline through 24 months
  Change from baseline in time to complete TUG
100-meter walk/run test (100MWT) | Baseline through 24 months
  Change from baseline in time to complete 100MWT

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | Baseline through 24 months
  Percent change from baseline in FVC
Muscle MRI | Baseline though 24 months
  Change from baseline in Fat fraction in thigh and leg skeletal muscles
Change from baseline in Activlim score | Baseline through 24 months
  Scale measuring level of limitation in performing daily activities (total score ranging from 0 to 44, with the lower score with highest limitation)

CONTACTS AND LOCATIONS:
Locations (3):
- Hopital Raymond Poincare, Garches, France
- Tunisia (2):
  - Hedi Chaker Hospital Child Neurology Department, Sfax
  - National Institute Mongi Ben Hmida of Neurology, Tunis